CLINICAL TRIAL: NCT00935311
Title: A Randomized, Multicenter, Single-blind, Placebo-controlled Study Comparing the Analgesic Efficacy and Safety of Hydrocodone/ Acetaminophen Extended-release Tablets and Hydrocodone/Acetaminophen (NORCO) to Placebo in Subjects With Acute Pain Following Third Molar Tooth Extraction
Brief Title: Hydrocodone/Acetaminophen for Acute Pain Following Third Molar Tooth Extraction
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AbbVie (prior sponsor, Abbott) (Industry)
Responsible Party: Sponsor
Organization: AbbVie (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: M11-063
Record Dates: First submitted 2009-06-29; First posted 2009-07-09 (Estimated); Results first posted 2014-03-07 (Estimated); Last update posted 2014-04-08 (Estimated); Status verified 2014-03

CONDITIONS: Pain
MeSH Terms: conditions — Pain | interventions — Hydrocodone

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- ABT-712 (Experimental): 1 dose of 1 ABT-712 extended-release tablet plus 1 placebo tablet, followed by 1 dose of 2 placebo tablets, administered once every 6 hours for 12 hours (for a total of 2 doses).
  Interventions: Drug: ABT-712 Extended-release; Drug: Placebo
- Hydrocodone/Acetaminophen (Active Comparator): 2 doses of 1 hydrocodone/acetaminophen immediate-release tablet plus 1 placebo tablet, administered once every 6 hours for 12 hours (for a total of 2 doses).
  Interventions: Drug: Hydrocodone/Acetaminophen Immediate-release; Drug: Placebo
- Placebo (Placebo Comparator): 2 doses of 2 placebo tablets, administered once every 6 hours for 12 hours (for a total of 2 doses).
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ABT-712 Extended-release — ABT-712 extended-release tablet
  Other Names: Hydrocodone/acetaminophen extended-release; Hydrocodone bitartrate and acetaminophen extended-release
  Arms: ABT-712
Drug: Hydrocodone/Acetaminophen Immediate-release — Hydrocodone/acetaminophen immediate-release tablet
  Arms: Hydrocodone/Acetaminophen
Drug: Placebo — Placebo tablet

SUMMARY:
The purpose of this study was to evaluate analgesic efficacy and safety of hydrocodone/acetaminophen compared to placebo in moderate to severe pain following molar extraction.

DETAILED DESCRIPTION:
Dosing started within 6 hours after completion of third molar extraction. Study drug was given once every 6 hours for 12 hours (for a total of 2 doses). Participants were randomized to receive placebo or active drug (either experimental drug or comparator). The total dose was the same for both groups receiving active drug, but was given as either 1 dose of extended-release tablets (experimental drug), or 2 doses of immediate-release tablets (active comparator).

ELIGIBILITY:
Inclusion Criteria:

* Subjects who are in general good health, experiencing moderate to severe pain after surgical extraction of 2 or more third molars and who are willing to remain confined until the morning after surgery for study procedures

Exclusion Criteria:

* Allergies to study medications
* History of multiple drug allergies
* Unable to stop excluded medications
* Clinically significant laboratory abnormalities at Screening
* Significant medical condition at Screening
* Women who are pregnant or breast feeding

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 122 (Actual)
Dates: Start 2009-06; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pedro Quintana Diez, MD, Study Director — AbbVie
Locations (3):
- United States (3):
  - Site Reference ID/Investigator# 20745, Austin, Texas
  - Site Reference ID/Investigator# 20743, San Marcos, Texas
  - Site Reference ID/Investigator# 20744, Salt Lake City, Utah

REFERENCES:
- See also: Related Info — http://rxabbvie.com

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | ABT-712 | Hydrocodone/Acetaminophen | Placebo
Started | 43 | 39 | 40
Completed | 43 | 39 | 40
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ABT-712 | Hydrocodone/Acetaminophen | Placebo | Total
Number analyzed (Participants) | 43 | 39 | 40 | 122
Age, Continuous [Mean (Standard Deviation); unit: years] | 22.1 (2.83) | 21.4 (3.20) | 23.0 (4.73) | 22.2 (3.70)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 23 | 28 | 73
  Male | 21 | 16 | 12 | 49

OUTCOME MEASURES:

1. Primary Outcome: Sum of Pain Intensity Difference (SPID) Using the Pain Intensity Visual Analog Scale (VAS)
Description: Participants assessed pain intensity on a 100 mm visual analogue scale (VAS) with 0 meaning "no pain" and 100 meaning the "worst pain imaginable". The SPID VAS score for 0 to 12 hours following initial study drug dose measured the cumulative pain intensity difference during treatment with higher mean SPID VAS scores indicating greater improvement from Baseline. The SPID score is a measure of the cumulative pain intensity difference during treatment and the area under the curve was estimated using the linear trapezoidal rule.
Time Frame: From time of first study drug administration to 12 hours following first study drug administration
Population: All randomized participants who received at least 1 dose of study drug.
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | ABT-712 | Hydrocodone/Acetaminophen | Placebo
Number analyzed (Participants) | 43 | 39 | 40
scores on a scale | 268.8 (44.29) | 230.9 (47.03) | 54.8 (46.19)

2. Secondary Outcome: TOTPAR (Total Pain Relief)
Description: TOTPAR was the time-interval weighted sum of pain relief. Pain relief was assessed by participants' responses to how their pain relief was compared with the pain they had just before receiving the first dose of study drug: no relief, a little relief, some relief, a lot of relief, or complete relief. Higher mean TOTPAR scores indicate better pain relief. The TOTPAR score is a measure of the cumulative pain intensity difference during treatment and the area under the curve was estimated using the linear trapezoidal rule.
Time Frame: From time of first study drug administration to 12 hours following first study drug administration
Population: All randomized participants who received at least 1 dose of study drug.
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | ABT-712 | Hydrocodone/Acetaminophen | Placebo
Number analyzed (Participants) | 43 | 39 | 40
scores on a scale | 18.0 (2.06) | 15.9 (2.16) | 10.5 (2.13)

3. Secondary Outcome: Time to First Rescue Medication
Description: The median time (minutes) from first dose of study drug to first use of analgesic rescue medication.
Time Frame: From time of first study drug administration to 12 hours following first study drug administration
Population: All randomized participants who received at least 1 dose of study drug.
Measure: Median (95% Confidence Interval); unit: minutes
Arm/Group | ABT-712 | Hydrocodone/Acetaminophen | Placebo
Number analyzed (Participants) | 43 | 39 | 40
minutes | 442.0 [196.0 to 612.0] | 205.0 [190.0 to 642.0] | 123.5 [104.0 to 153.0]

4. Secondary Outcome: Participants With Adverse Events (AEs)
Description: An adverse event (AE) is defined as any untoward medical occurrence in a participant, which does not necessarily have a causal relationship with treatment. If an adverse event meets any of the following criteria, it is considered a serious adverse event (SAE): results in death or is life-threatening, results in admission or prolongation of hospitalization, results in congenital anomaly or persistent or significant disability/incapacity, or is an important medical event requiring medical or surgical intervention to prevent serious outcome. AEs were categorized by severity (mild, moderate, severe) and relationship to treatment (probably, possibly, probably not, not related). Please see Adverse Events section below for more details.
Time Frame: AEs were recorded from study drug administration until 30 days following discontinuation of study drug (total 30 days); SAEs were recorded from the time informed consent was obtained until 30 days following discontinuation of study drug (total 51 days).
Population: All randomized participants who received at least 1 dose of study drug.
Measure: Number; unit: participants
Arm/Group | ABT-712 | Hydrocodone/Acetaminophen | Placebo
Number analyzed (Participants) | 43 | 39 | 40
participants
  Any AE | 14 | 12 | 14
  Any AE at least "possibly" drug related | 5 | 8 | 4
  Any AE at least "probably not" drug related | 9 | 4 | 10
  Any "severe" AE | 1 | 0 | 2
  Any SAE | 0 | 0 | 0
  Any AE leading to discontinuation of study drug | 0 | 0 | 0
  Any AE leading to death | 0 | 0 | 0
  Death | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: AEs were recorded from study drug administration until 30 days following discontinuation of study drug (total 30 days); SAEs were recorded from the time informed consent was obtained until 30 days following discontinuation of study drug (total 51 days).
Arm/Group | ABT-712 | Hydrocodone/Acetaminophen | Placebo
Serious Adverse Events (participants affected / at risk) | 0/43 | 0/39 | 0/40
Other Adverse Events (participants affected / at risk) | 11/43 | 10/39 | 13/40
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | ABT-712 (N=43) | Hydrocodone/Acetaminophen (N=39) | Placebo (N=40)
DIARRHOEA (Gastrointestinal disorders) | 0 | 0 | 2
NAUSEA (Gastrointestinal disorders) | 7 | 7 | 2
VOMITING (Gastrointestinal disorders) | 1 | 2 | 2
CHILLS (General disorders) | 0 | 0 | 2
DIZZINESS (Nervous system disorders) | 1 | 5 | 3
HEADACHE (Nervous system disorders) | 5 | 0 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.